CLINICAL TRIAL: NCT06265922
Title: Effect of Cerebellar Repetitive Transcranial Magnetic Stimulation on Coordination in Patients with Multiple Sclerosis
Brief Title: Cerebellar RTMS in Patients with Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Zayed Abd Elraheem Mohamed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003937
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Patients with Multiple Sclerosis
Keywords: Patients with Multiple Sclerosis; Coordination; Transcranial magnetic stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant masking as patients will be divided into two groups High frequecy cerebellar repetitive transcranial magnetic stimulation and Sham repetitive transcranial magnetic stimulation by placing the coil in perpendicular way away from the cerebellum.
  Care provider masking as the physical therapist treating patients will be blind from the application of repetitive transcranial magnetic stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High frequency cerebellar repetitive transcranial magnetic stimulation (Active Comparator): Twenty patients will be treated by high frequency repetitive transcranial magnetic stimulation (Hf-rTMS) targeting the cerebellum beside a tailored physical therapy program designed for the ataxic manifestation The protocol of rTMS included 6 sessions over 2 weeks. MagPro R20 device will be applied over midline of cerebellum using circular coil. Ten repetition rate in 40 trains with one inter train interval will be applied two times within the same session, 5 minutes rest in between Tailored physiotherapy program for ataxic manifestation will be applied for 10 days in the same 2 weeks
  Interventions: Device: High frequency repetitive transcranial magnetic stimulation
- Sham cerebellar repetitive transcranial magnetic stimulation (Sham Comparator): Twenty patients will be treated by sham cerebellar rTMS with the same parameters, same duration 6 sessions over 2 weeks except the coil will not be on the middle of the cerebellum instead it will be perpendicular away from it.
  But the program of physiotherapy is the same
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: High frequency repetitive transcranial magnetic stimulation — High frequency repetitive transcranial magnetic stimulation will be applied over mid line of cerebellum using circular coil. Ten repetition rate (frequency) in 40 trains with one intertrain interval will be applied for three times a week for two weeks.
  Other Names: Hf-rTMS
  Arms: High frequency cerebellar repetitive transcranial magnetic stimulation
Device: Sham repetitive transcranial magnetic stimulation — Sham repetitive transcranial magnetic stimulation will be applied Perpendicular away from the cerebellum using the same circular coil. The same parameters will be used with the same duration also numbers of sessions are the same like the active comparator group to assure the patients blindness
  Arms: Sham cerebellar repetitive transcranial magnetic stimulation

SUMMARY:
To determine the efficacy of high frequency cerebellar repetitive transcranial magnetic stimulation on coordination in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Forty patients with multiple sclerosis suffering from ataxia less than five in EDSS score will be recruited from the outpatient clinic at Faculty of Physical Therapy as well as Kasr Al-Ainy Multiple Sclerosis unit (KAMSU), Cairo University. The study will be applied during the remission period. Patients will be assessed by Biodex balance system, Berg balance scale, Four square step test and Nine-Hole Peg Test to investigate coordination in both equilibrium and non-equilibrium. Patient will be divided into two groups.The study group will be treated by High frequecy cerebellar repetitive transcranial magnetic stimulation besides a tailored physiotherapy program, while the control group will be treated by Sham cerebellar repetitive transcranial magnetic stimulation with a tailored physiotherapy program as well. The treatment duration for each patient will take weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS (relapsing, remitting and secondary progressive) patients
* Patients who are medically stable and Free from relapses three months before
* Ambulant patients without an assistive device and score less than 5 on the Kurtzke Expanded Disability Status Scale (EDSS)
* Patients receiving their disease modifying drugs but no medication changing during the previous three months.
* Patients who had MRI evidence of lesions in the cerebellum or in the cerebellar pedunculi.
* Right handed patients.
* Severity of ataxia range from 4 to 10 according to scale of assessment and rating ataxia (SARA).
* Did not apply cerebellar transcranial magnetic stimulation before.

Exclusion Criteria:

* Any other neurological deficits or orthopedics abnormalities.
* Ataxic manifestations for other cause rather than Multiple Sclerosis.
* Other neurological manifestations (e.g. spasticity, visual loss)
* Secondary musculoskeletal complication such as contractures or deformities. Cardiovascular, pulmonary, hepatic, renal, hemopoietic and thyroid diseases.
* Pregnant women.
* Addicted individuals.
* Previous surgeries in the brain.
* Any magnetic or metallic devices implanted (like cochlear implants) .
* Psychotic deficits or history of epileptic seizures.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Biodex balance system | 2 weeks after end of treatment
  Change of balance and stability index from baseline to 2 weeks after the beginning of intervention (when the score decreases, this means good)

SECONDARY OUTCOMES:
Berg balance scale | 2 weeks after end of treatment
  Change of the balance score from baseline to two weeks after the beginning of the intervention ( the scale consists of 14 item. Minimum score for each item is 0 and maximum score is 4, to record the patient the summation of the 14 item is counted. And if the score is increasing this means good)
Nine-Hole Peg Test (9-HPT) | 2 weeks after end of treatment
  Change of manual dexterity of both the dominant and non dominant hand from baseline to 2 weeks after the beginning of intervention
Four square step test (FSST) | 2 weeks after end of treatment
  Change of dynamic balance and coordination from baseline to 2 weeks after the beginning of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Dokki, Egypt

REFERENCES:
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Aloizou AM, Pateraki G, Anargyros K, Siokas V, Bakirtzis C, Liampas I, Nousia A, Nasios G, Sgantzos M, Peristeri E, Dardiotis E. Transcranial magnetic stimulation (TMS) and repetitive TMS in multiple sclerosis. Rev Neurosci. 2021 Feb 25;32(7):723-736. doi: 10.1515/revneuro-2020-0140. Print 2021 Nov 25. PMID 33641274
- [Background] Somaa FA, de Graaf TA, Sack AT. Transcranial Magnetic Stimulation in the Treatment of Neurological Diseases. Front Neurol. 2022 May 20;13:793253. doi: 10.3389/fneur.2022.793253. eCollection 2022. PMID 35669870
- [Derived] Mohamed HZA, Elwishy AA, Shalaby NM, Shehata HSM, Ali AS. Cerebellar repetitive transcranial magnetic stimulation combined with physiotherapy for balance in people with multiple sclerosis: A randomized controlled trial with six-week follow-up. Mult Scler Relat Disord. 2025 Oct;102:106610. doi: 10.1016/j.msard.2025.106610. Epub 2025 Jul 9. PMID 40664092